CLINICAL TRIAL: NCT01307384
Title: Prospective Post Market Clinical Follow-Up Study of the Continuum Metal on Polyethylene Acetabular System
Brief Title: Zimmer Continuum Metal on Polyethylene (MoP) PostMarket Clinical Followup (PMCF) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2010-02H
Record Dates: First submitted 2011-02-25; First posted 2011-03-02 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Avascular Necrosis; Osteoarthritis; Inflammatory Arthritis; Post-traumatic Arthritis; Rheumatoid Arthritis
Keywords: Total Hip Arthroplasty; Total Hip Replacement (THR); Primary Hip Arthroplasty; THA; THR
MeSH Terms: conditions — Osteonecrosis; Osteoarthritis; Arthritis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Continuum Acetabular System: Patients receiving primary hip arthroplasty using the Continuum Metal on Polyethylene Acetabular System
  Interventions: Device: Continuum Metal on Polyethylene Acetabular System

INTERVENTIONS:
Device: Continuum Metal on Polyethylene Acetabular System — Used in primary hip arthroplasty
  Other Names: Total Hip Replacement, Total Hip Arthroplasty, Primary Hip

SUMMARY:
This is a prospective, multi-center, non-randomized, non-controlled study designed to obtain survival and outcome data on the Continuum Metal on Polyethylene Acetabular System when used in primary total hip arthroplasty.

DETAILED DESCRIPTION:
The safety and performance of the Continuum Metal on Polyethylene Acetabular System will be confirmed by the assessment of survival and outcome data. Assessments will include standard scoring systems, radiographs and adverse event records. Data will be used to monitor pain, mobility, and survivorship of the Continuum Metal on Polyethylene Acetabular system in primary total hip arthroplasty. Metal ion (cobalt, chromium and titanium) and renal function (BUN, Creatinine and GFR) levels will be analyzed for a subset of the enrolled study subjects.

ELIGIBILITY:
Inclusion Criteria

* Patient is 18 to 75 years of age, inclusive.
* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral (simultaneous or staged) total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Avascular necrosis (AVN)
  * Osteoarthritis
  * Inflammatory arthritis (i.e., Rheumatoid arthritis)
  * Post-traumatic arthritis
* Patient has no history of previous prosthetic replacement device of any type, including surface replacement arthroplasty, endoprosthesis, etc. of the affected hip joint(s).
* Patient has moderate, marked or disabling pain.
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the IRB approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant
* The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure or complications in postoperative care.
* The patient has a neurologic condition in the ipsilateral or contralateral limb which affects lower limb function.
* The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give consent or to comply with the follow-up program.
* The patient has received an investigational drug or device within the previous 6 months.
* The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
* The patient has insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e., osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be used to assess the presence of adequate bone stock.
* The patient has osteoradionecrosis in the affected hip joint.
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials.
* The patient has known local bone tumors and/or cysts in the operative hip.
* The patient has a Body Mass Index (BMI) > 40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from surgeons medical practice who are candidates for primary hip arthroplasty.
  The study population will be comprised of 300 males and females who require primary total hip arthroplasty. Subjects will be enrolled at up to 7 clinical sites. Subjects must be geographically accessible throughout the study and be willing and able to attend required follow-up appointments. Candidates who express interest in study participation will be offered informed consent, and eligibility will be determined based upon the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 6 weeks, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year, and 10 year
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method.
Safety / Adverse Events | Surgery, 6 weeks, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year, and 10 year
  Safety will be evaluated by monitoring the frequency and incidence of device related adverse events or unanticipated adverse device effects in investigational subjects.

SECONDARY OUTCOMES:
Pain and Function / HHS | 6 weeks, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year, and 10 year
  Pain and function will be measured using the Harris Hip Score self assessment.
Pain and Function / OHS | 6 weeks, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year, and 10 year
  Pain and function will be measured using the Oxford Hip Score self assessment.
Health Status / SF-12 | 6 weeks, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year, and 10 year
  Health status will be measured using the SF-12 self assessment.
Health Status / Radiographic Parameters | 6 weeks, 6 months, 1 year, 2 year, 3 year, 5 year, 7 year, and 10 year
  X-rays will be evaluated for acetabular cup angle, acetabular cup migration, femoral stem position, femoral stem subsidence and femoral stem shift.

OTHER OUTCOMES:
Metal Ion / Cobalt | Pre-operatively and at 6 months, 1 year, 2 year and 5 years
  Blood specimens analyzed for a subset of all enrolled study subjects to use as a comparator to blood levels in patients being studied under a separate clinical protocol. Adverse events reported for levels outside of normal range.
Metal Ion / Chromium | Pre-operatively and at 6 months, 1 year, 2 year and 5 years
  Blood specimens analyzed for a subset of all enrolled study subjects to use as a comparator to blood levels in patients being studied under a separate clinical protocol. Adverse events reported for levels outside of normal range.
Metal Ion / Titanium | Pre-operatively and at 6 months, 1 year, 2 year and 5 years
  Blood specimens analyzed for a subset of all enrolled study subjects to use as a comparator to blood levels in patients being studied under a separate clinical protocol. Adverse events reported for levels outside of normal range.
Renal Function / BUN | Pre-operatively and at 6 months, 1 year, 2 year and 5 years
  Blood specimens analyzed for a subset of all enrolled study subjects to use as a comparator to blood levels in patients being studied under a separate clinical protocol. Adverse events reported for levels outside of normal range.
Renal Function / Creatinine | Pre-operatively and at 6 months, 1 year, 2 year and 5 years
  Blood specimens analyzed for a subset of all enrolled study subjects to use as a comparator to blood levels in patients being studied under a separate clinical protocol. Adverse events reported for levels outside of normal range.
Renal Function / GFR | Pre-operatively and at 6 months, 1 year, 2 year and 5 years
  Blood specimens analyzed for a subset of all enrolled study subjects to use as a comparator to blood levels in patients being studied under a separate clinical protocol. Adverse events reported for levels outside of normal range.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - Sah Orthopaedic Associates, Fremont, California
  - Denver Health Medical Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No